CLINICAL TRIAL: NCT00670332
Title: Prognostic Assessment of Contrast Echocardiography (PACE Study): An Observational Follow-up Study of Patients With Chest Pain Evaluated With AI-700 Contrast Echocardiography
Brief Title: Prognostic Assessment of Contrast Echocardiography (PACE Study)
Acronym: PACE
Status: Terminated | Type: Observational
Sponsor: Acusphere (Industry)
Responsible Party: Johh F. Cavanaugh, Acusphere
Other Study IDs: AI-700-36
Expanded Access: Available
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Last update posted 2008-05-01 (Estimated); Status verified 2008-04

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; echocardiography; cardiac imaging; heart disease; ultrasound contrast agent; prognosis
MeSH Terms: conditions — Coronary Artery Disease; Heart Diseases

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
This study will demonstrate whether patients with prognostically-significant myocardial abnormalities detected with AI-700 contrast ECHO have a rate of cardiac death or MI that is higher than that of patients with normal AI-700 contrast ECHO.

DETAILED DESCRIPTION:
This observational study will investigate the ability of AI-700 contrast ECHO to predict risk of future cardiovascular events occurring in patients who had a recent history of chest pain at the time of ECHO evaluation. Eligible patients were enrolled in either AI-700-32 or AI-700-33, which are completed Phase 3 international, multicenter, open-label, dual-injection studies of the myocardial imaging capabilities and safety of AI-700 administered intravenously in patients with chest pain. In the course of these Phase 3 studies, patients were evaluated with AI-700 contrast ECHO. In addition, eligible patients were to have had an evaluable pharmacologic stress-induced AI-700 ECHO assessment as part of AI-700-32 or AI-700-33.

ELIGIBILITY:
Eligible patients were enrolled in either AI-700-32 or AI-700-33.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This observational study will enroll up to 773 patients who participated in either AI-700-32 or AI-700-33 and who were evaluated with AI-700 contrast ECHO at rest and at pharmacologic-induced stress. Approximately 28 international study centers will participate. At the time of AI-700 contrast ECHO (defined as the index date), the patients were to have had a recent history of chest pain and were to meet all eligibility criteria. Chest pain (angina) was defined as either:
  * typical chest pain: 1) substernal chest discomfort with a characteristic quality and duration that is 2) provoked by exertion or emotional stress and 3) relieved by rest or nitroglycerin, or
  * atypical chest pain (angina) that meets 2 of the 3 typical chest pain characteristics.
Sampling Method: Non-Probability Sample
Enrollment: 773 (Estimated)
Dates: Start 2007-07

PRIMARY OUTCOMES:
The primary outcome variable is the time to first occurrence of the composite outcome (death or confirmed non fatal MI). | The time between AI 700 ECHO and outcomes data collection will be ≥12 months with an expected average follow-up period of 24 months

SECONDARY OUTCOMES:
Certain secondary analyses will include revascularizations and CHF. | The time between AI 700 ECHO and outcomes data collection will be ≥12 months with an expected average follow-up period of 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Acusphere, Watertown, Massachusetts, United States